CLINICAL TRIAL: NCT01726738
Title: LCCC 1128: Open Label Phase II Trial of the BRAF Inhibitor (Dabrafenib) and the MEK Inhibitor (Trametinib) in Unresectable Stage III and Stage IV BRAF Mutant Melanoma; Correlation of Resistance With the Kinome and Functional Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1128
Record Dates: First submitted 2012-11-08; First posted 2012-11-15 (Estimated); Results first posted 2020-09-07 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-09

CONDITIONS: Stage III Melanoma; Stage IV Melanoma; Unresectable Melanoma; BRAF Mutant Melanoma
Keywords: Melanoma; Stage III; Stage IV; Unresectable; BRAF Mutant; Dabrafenib; Trametinib; Kinome; Resistance; Sequencing; Mutations; Kinases; Mechanism
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BRAF (dabrafenib) and MEK (trametinib) inhibitors (Experimental): Patients will receive the BRAF inhibitor dabrafenib and MEK inhibitor trametinib orally at the RP2D determined in the Phase I/II study (BRF113220): trametinib 2mg QD and dabrafenib 150 mg BID on a continuous basis. A cycle will be defined as 3 weeks in duration. Cycles will be repeated until disease progression (clinical or radiological). Patients may remain on treatment after progression (at the discretion of the investigator) as long as they are still experiencing clinical benefit.
  Interventions: Drug: BRAF inhibitor dabrafenib and MEK inhibitor trametinib

INTERVENTIONS:
Drug: BRAF inhibitor dabrafenib and MEK inhibitor trametinib — Patients will receive the BRAF inhibitor dabrafenib and MEK inhibitor trametinib orally at the RP2D determined in the Phase I/II study (BRF113220): trametinib 2mg QD and dabrafenib 150 mg BID on a continuous basis. A cycle will be defined as 3 weeks in duration. Cycles will be repeated until disease progression (clinical or radiological). Patients may remain on treatment after progression (at the discretion of the investigator) as long as they are still experiencing clinical benefit.
  Other Names: BRAF Inhibitor Dabrafenib GSK2118436; MEK Inhibitor Trametinib GSK1120212

SUMMARY:
This phase II study in 20 patients with BRAFV600E mutant, unresectable stage III/IV melanoma is designed to explore the mechanisms by which tumors acquire resistance to the combination of a BRAF inhibitor (dabrafenib) and MEK inhibitor (trametinib). Tissue will be collected at baseline and at progression.If a subject is removed from the study for one of a variety of reasons including, but not limited to, an inability to tolerate the combination of dabrafenib and trametinib, a need to receive other therapy or completion of 3-years of study treatment without progression, and the subject later receives, as part of his/her standard of care, the combination of dabrafenib and trametinib and progresses on the standard of care regimen, then the subject may be contacted by the treating physician to be put back on to the LCCC 1128 protocol and have a progression biopsy at this progression time point. Markers of resistance will be explored by performing near kinome-wide profiling on tumor samples, and in patients who co-enroll in institutional protocol LCCC1108, by sequencing tumors using NextGen DNA sequencing technology. Overall response rate and duration to this combination will also be assessed.

DETAILED DESCRIPTION:
The present phase II study in 20 patients with BRAFV600E mutant, unresectable stage III/IV melanoma is designed to explore the mechanisms by which tumors acquire resistance to the combination of BRAF and MEK inhibition. Overall response rate and duration to this combination will also be assessed.

Tissue will be collected at baseline and at progression (clinical or radiological). Patients may remain on treatment after progression (at the discretion of the investigator) as long as they are still experiencing clinical benefit. We anticipate that up to 50% of patients may continue on therapy post-progression for 2-8 weeks.

BRF113220, the phase I/II trial of the BRAF inhibitor dabrafenib in combination with the MEK inhibitor trametinib is ongoing in metastatic melanoma to establish the safety of this combination, and to determine the recommended phase 2 doses (RP2D) for each agent. Expansion cohorts at the RP2D for these drugs in combination were included in the phase I to characterize the safety in more detail, and to explore the efficacy of this combination. The combination was well tolerated as described in section 1.5, with decreased frequency of rash compared to either agent alone and with just 1 report of cutaneous SCC.

This proposed study will utilize the RP2D determined in the Phase I/II study: trametinib 2mg QD and dabrafenib 150 mg BID. Despite a very promising overall response rate of 81%, these patients will also likely go on to develop resistance as a result of new resistance mutations, and given the cooperative signaling network of kinases that sense inhibition of key nodal kinases and induce compensatory responses that offset pharmacological intervention. The study objectives are as follows: Objectives Primary Objective To identify kinases that are differentially expressed pre- and post-treatment with BRAF (dabrafenib) and MEK (trametinib) inhibitors, and to determine a kinome signature predictive of resistance to BRAF/MEK inhibition in stage III/IV melanoma Secondary Objectives To explore whether resistance to BRAF and MEK inhibition is associated with new functional mutations in the approximately 150 oncogenes / tumor suppressor genes that are assessed in more than 10% of the tumors (using NextGen DNA sequencing technology) in the subset of patients who co-enroll in LCCC1108, with particular focus on one of five established resistance genes (BRAF, NRAS, MEK1, MAP3K8 or COT, and PTEN) To determine the overall response rate (ORR: complete response + partial response) as measured via RECISTv1.1 To estimate the duration of ORR as measured via RECISTv1.1 To estimate progression-free survival (PFS) as defined by RECISTv1.1 To estimate the rate of overall survival (OS) at 1 year from day 1 of treatment

Primary Endpoint Kinome signature pathway will be based on comparison of kinome expression from pre- and post-treatment biopsies using Multiplexed Inhibitor Beads (MIBs) coupled with mass spectrometry.

ELIGIBILITY:
Main Study Inclusion Criteria:

Subject must meet all of the inclusion criteria to participate in this study:

Age ≥18 years Signed written informed consent Histologically confirmed V600E or V600K BRAF mutant melanoma Unresectable Stage III/IV melanoma ECOG PS 0-2

Normal organ function as defined by the following:

* Absolute neutrophil count >1.2 × 109/L
* Hemoglobin >9 g/dL, platelets >75 × 109/L
* PT/INR and PTT ≤1.5 x ULN (Note: subjects receiving anticoagulation treatment may enroll with INR established within the therapeutic range prior to D1 of treatment)
* Albumin >2.5 g/dL
* Total bilirubin <1.5 x ULN (patients with elevated bilirubin due to Gilbert's disease will not be excluded)
* AST and ALT < 2.5× ULN
* CrCl ≥50mL/min per Cockcroft-Gault Prior anti-cancer treatment related toxicities except alopecia and lab values as outlined in the criterion above must be less than or equal to Grade 1 as per CTCAEv4 Willing to undergo biopsy for research purposes only Females of child-bearing potential: willing to use two forms of effective contraception, and to continue use for 16 weeks post last dose of study medication. Effective contraception is defined as any medically recommended method (or combination of methods) as per standard of care, including abstinence. Females of non-childbearing potential are those who are postmenopausal (defined as greater than 1 year without menses with appropriate clinical profile, e.g., age appropriate: >45 years in the absence of hormone replacement therapy (HRT). In questionable cases, the subject must have a follicle stimulating hormone (FSH) value >40 mIU/mL and an estradiol value <40pg/mL (<140 pmol/L); or who have had a bilateral tubal ligation or tubal occlusion, bilateral oophorectomy, or hysterectomy. Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception as described from D1 of treatment, throughout the treatment period, and for 16 weeks after the last dose of study treatment. If a subject becomes pregnant during the treatment period of the study, the study treatments should be stopped immediately.

In women of child-bearing potential, negative serum pregnancy test within 48 hours prior to day 1 of study treatment and agree to use effective contraception. Effective contraception is defined as: (a) an intrauterine device with a documented failure rate of less than 1% per year. (b) male partner sterilization prior to the female subject's entry, and this male is the sole sexual partner for that female. (c) complete abstinence from sexual intercourse for 14 days prior to enrollment throughout study treatment, and for at least 4 months after the last dose of study treatment. Abstinence is only acceptable when in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar ovulation, symptothermal, post-ovulation methods, etc) and withdrawal are not acceptable methods of contraception. (d) double- barrier contraception: condom and occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/cream/suppository). Note: hormonal based methods (e.g. oral contraceptives) are not permitted.

Female subjects who are lactating must discontinue nursing prior to the first dose of study treatment and must refrain from nursing throughout the treatment period and for 4 months following the last dose of study treatment Measurable disease as defined by RECIST v1.1 Able to swallow and retain oral medication Left ventricular ejection fraction by ECHO ≥ institutional lower limit of normal

Main Study Exclusion Criteria:

Any subject meeting any of the following exclusion criteria at baseline will be ineligible for study participation:

Patients with a history of a prior malignancy are excluded unless they have been disease free for 3 or more years or unless they have a completely resected non-melanoma skin cancer, and/or subjects with indolent second malignancies.

History of malignancy with confirmed activating RAS mutation at any time. Note: Prospective RAS testing is not required. However, if the results of previous RAS testing are known, they must be used in assessing eligibility.

Prior treatment with a BRAF inhibitor (including but not limited to dabrafenib (GSK2118436), vemurafenib, and LX281/BMS-908662) or a MEK inhibitor (including but not limited to trametinib (GSK1120212), AZD6244, and RDEA119); NOTE: There is no limit to the number of other prior therapies, and patients may be previously untreated.

Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study drug, or excipients or to dimethyl sulfoxide (DMSO).

Active GI or intracranial hemorrhage

History or evidence of cardiovascular risk including any of the following:

* QTc ≥ 480 msec;
* History or evidence of current clinically significant uncontrolled arrhythmias;

  o Exception: Subjects with controlled atrial fibrillation for >30 days prior to D1 of study treatment are eligible.
* History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to study entry;
* Patients with history of hypertension should have hypertension adequately controlled (BP<140/90) with appropriate anti-hypertensive therapy or diet prior to study entry;
* Patients with intra-cardiac defibrillators or permanent pacemakers;
* Known cardiac metastases;
* Abnormal cardiac valve morphology (≥grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study.

History of known glucose-6-phosphate dehydrogenase (G6PD) deficiency

Brain metastases are excluded unless:

* All known lesions were previously treated with surgery or stereotactic surgery (whole-brain radiation is not allowed unless given after definitive treatment with surgery or stereotactic surgery), AND
* Brain lesion(s), if still present, must be confirmed stable (i.e., no increase in lesion size) for ≥ 12 weeks prior to D1 of study treatment (stability must be confirmed with two consecutive magnetic resonance image (MRI) or computed tomography (CT) scans with contrast, AND
* Asymptomatic with no corticosteroid requirements for ≥ 4 weeks prior to D1 of study treatment, AND
* Treatment with any CYP enzyme inducing anticonvulsants occurred < 4 weeks prior to D1 of study treatment

NOTE: if study subject has history of brain metastasis, but currently has no evidence of disease in brain (NED), confirmation by two consecutive scans separated by ≥6 weeks prior to D1 of treatment is required.

Pulmonary embolism on active therapy History of interstitial lung disease or pneumonitis Known HIV, Hepatitis B or C infection (with the exception of chronic or cleared HBV and HCV infection which will be allowed provided the following tests are done at screening: viral hepatitis serology, Hepatitis B surface antigen and Hepatitis B core antibody (IgM) and/or Hepatitis C RNA) Currently active GI disease, or prior surgery that may affect ability to absorb oral medications

History or current evidence/risk of retinal vein occlusion (RVO) or retinal pigment epithelial detachment (RPED):

* Predisposing factors to RVO or RPED (e.g. uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as hypertension, diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes)
* Visible retinal pathology as assessed by ophthalmic exam that is considered a risk factor for RVO or CSR such as:

  * Evidence of new optic disc cupping
  * Evidence of new visual field defects
  * Intraocular pressure > 21 mm Hg Currently receiving cancer therapy (chemotherapy, radiotherapy, immunotherapy, or biologic therapy) NOTE: palliative radiation therapy is permitted for non-target lesions that are either new or present at baseline provided total dose does not exceed 30 Gy. However, radiation skin injury has been reported with concurrent use of dabrafenib and radiation. To reduce this risk, it is recommended that dabrafenib be held for seven days before and two days after radiation in subjects receiving dabrafenib in combination with trametinib when palliative radiation is prescribed.

Use of other prohibited medications within 5 half-lives or 14 days prior to the first dose of study drugs or requires any of these medications while receiving medication on this study Pregnant or lactating female

Inclusion Criteria for Off-Study Subjects to Receive Progression Biopsy

Currently progressing on Trametinib/Deabrafenib Combination Therapy

Willing to undergo biopsy for research purposes only.

Tumor amenable to research biopsy.

Signed written informed consent to have a progression biopsy performed on the LCCC 1128 protocol.

Previously enrolled on the LCCC 1128 study and did not have a progression biopsy previously performed while on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-04-04 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2020-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Lee, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Lineberger Comprehensive Cancer Center, UNC Chapel Hill, NC — http://www.unclineberger.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 17 participants were recruited from University of North Carolina Hospitals (Chapel Hill, NC) between January 2013 and July 2016
Pre-assignment Details: In addition to the 17 patients who were enrolled and participated in the trial, 6 additional patients consented, but were found to be ineligible and 1 additional patient withdrew consent prior to starting the study.
Groups:
- BRAF (Dabrafenib) and MEK (Trametinib) Inhibitors: BRAF inhibitor dabrafenib and MEK inhibitor trametinib: Patients received the BRAF inhibitor dabrafenib and MEK inhibitor trametinib orally at the Recommend Phase 2 Dose (RP2D) determined in the Phase I/II study (BRF113220): trametinib 2mg once a day (QD) and dabrafenib 150 mg twice a day (BID) on a continuous basis. A cycle is defined as 3 weeks in duration. Cycles were repeated until disease progression (clinical or radiological). Patients could remain on treatment after progression (at the discretion of the investigator) as long as they are still experiencing clinical benefit.
Period: Overall Study
Arm/Group | BRAF (Dabrafenib) and MEK (Trametinib) Inhibitors
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- BRAF (Dabrafenib) and MEK (Trametinib) Inhibitors: BRAF inhibitor dabrafenib and MEK inhibitor trametinib: Patients received the BRAF inhibitor dabrafenib and MEK inhibitor trametinib orally at the RP2D determined in the Phase I/II study (BRF113220): trametinib 2mg QD and dabrafenib 150 mg BID on a continuous basis. A cycle is defined as 3 weeks in duration. Cycles were repeated until disease progression (clinical or radiological). Patients could remain on treatment after progression (at the discretion of the investigator) as long as they are still experiencing clinical benefit.
Arm/Group | BRAF (Dabrafenib) and MEK (Trametinib) Inhibitors
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 54 [36 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Kinase Expression
Description: The primary outcome of this study is to identify kinases that are differentially expressed pre- and post-treatment with BRAF (dabrafenib) and MEK (trametinib) inhibitors. The kinases will be profiled using Multiplexed Inhibitor Beads (MIBs) coupled with mass spectrometry (MS) and reported as a sum of the Log 2 Fold Change between baseline and one year post treatment across all patients
Time Frame: Baseline and One year post treatment
Population: Progression samples were not available for 7 participants; 3 additional participants did not have samples that were evaluable by MIB/MS
Measure: Number; unit: Sum Log 2 Fold Change Kinase Expression
Arm/Group | BRAF (Dabrafenib) and MEK (Trametinib) Inhibitors
Number analyzed (Participants) | 7
Sum Log 2 Fold Change Kinase Expression
  RIPK2 | -20.87259
  PTK6 | -19.64376
  BRAF | -16.41738
  CDK1 | -12.5401
  PAK4 | -12.31239
  LIMK1 | -12.38811
  EIF2AK2 | -12.51229
  AURKA | -10.87395
  PI4K2B | -7.66173
  PKMYT1 | -11.3527
  MAP4K3 | -9.8909
  WEE1 | -9.61838
  TEC | -10.15407
  CSNK1D | -9.57122
  EPHA4 | -9.5134
  AURKB | -5.70255
  ZAK | -9.14964
  LIMK2 | -7.86008
  ADCK4 | -8.56373
  NME4 | -5.34905

2. Primary Outcome: Kinome Signature Predictive of Resistance
Description: Prediction analysis of microarrays (PAM) based on nearest shrunken centroid will also be carried out to identify a subset of kinases that predicts resistance to BRAF+MEK inhibition.
Time Frame: One year post treatment
Measure: Number; unit: predictive kinase signatures
Arm/Group | BRAF (Dabrafenib) and MEK (Trametinib) Inhibitors
Number analyzed (Participants) | 7
predictive kinase signatures | 0

3. Secondary Outcome: BRAF and MEK Inhibition Associated With New Functional Mutations in the Approximately 150 Oncogenes
Description: The secondary outcome measure is to explore whether resistance to BRAF and MEK inhibition is associated with new functional mutations in the approximately 150 oncogenes / tumor suppressor genes that are assessed in more than 10% of the tumors (using Next Generation (NextGen) DNA sequencing technology) in the subset of patients who co-enroll in a correlative study, with particular focus on one of five established resistance genes (BRAF, NRAS, MEK1, Mitogen-Activated Protein Kinase Kinase Kinase 8 (MAP3K8) or Cancer Osaka Thyroid (COT), and PTEN).
Time Frame: One year
Population: as for outcome 1
Measure: Number; unit: Functional mutation predictors
Arm/Group | BRAF (Dabrafenib) and MEK (Trametinib) Inhibitors
Number analyzed (Participants) | 7
Functional mutation predictors | 0

4. Secondary Outcome: Overall Response Rate (ORR)
Description: To determine the disease overall response rate (ORR: complete response (CR) + partial response (PR)/total number of patients) as measured radiographically via Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions. CR is defined as the disappearance of all target lesions; PR is a >=30% decrease in the sum of the longest diameter of target lesions
Time Frame: One year post treatment
Measure: Number (95% Confidence Interval); unit: percentage of patients with response
Arm/Group | BRAF (Dabrafenib) and MEK (Trametinib) Inhibitors
Number analyzed (Participants) | 17
percentage of patients with response | 76 [50 to 93]

5. Secondary Outcome: Duration of Overall Response
Description: Duration of overall response is defined as the time from documentation of response (Complete or Partial) to time of disease progression or death. Response was measured radiographically using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions. Complete Response is defined as the disappearance of all target lesions; Partial Response as a >=30% decrease in the sum of the longest diameter of target lesions, and Progressive Disease as a 20% increase in the sum of the longest diameter of target lesions or the appearance of new lesions.
Time Frame: One year post treatment
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | BRAF (Dabrafenib) and MEK (Trametinib) Inhibitors
Number analyzed (Participants) | 17
Months | 13 [1.4 to 22]

6. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from Day 1 of protocol treatment to the date of progression as measured radiographically using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) or to the date of death. Per RECIST, Progressive Disease as a 20% increase in the sum of the longest diameter of target lesions or the appearance of new lesions.
Time Frame: One year post treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BRAF (Dabrafenib) and MEK (Trametinib) Inhibitors
Number analyzed (Participants) | 17
Months | 17 [4.1 to 25.4]

7. Secondary Outcome: Rate of Overall Survival (OS) at 12 Months
Description: The rate of overall survival is defined as the percentage of patients still alive at one year from Day 1 of protocol treatment
Time Frame: One year post treatment
Measure: Number (95% Confidence Interval); unit: percentage of patients alive at 1 year
Arm/Group | BRAF (Dabrafenib) and MEK (Trametinib) Inhibitors
Number analyzed (Participants) | 17
percentage of patients alive at 1 year | 70 [42 to 86]

ADVERSE EVENTS:
Time Frame: From start of treatment through 30 days after end of treatment
Arm/Group | BRAF (Dabrafenib) and MEK (Trametinib) Inhibitors
All-Cause Mortality (participants affected / at risk) | 6/17
Serious Adverse Events (participants affected / at risk) | 11/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BRAF (Dabrafenib) and MEK (Trametinib) Inhibitors (N=17)
Alanine Aminotransferase Increased (Investigations) | 1
Aspartate Aminotransferase Increased (Investigations) | 1
Diarrhea (Gastrointestinal disorders) | 1
Endocrine Disorders - Other, Specify (Endocrine disorders) | 1
Fatigue (General disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 2
Flu Like Symptoms (General disorders) | 1
Gastrointestinal Disorders - Other, Specify (Gastrointestinal disorders) | 1
General Disorders And Administration Site Conditions - Other, Specify (General disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Intracranial Hemorrhage (Nervous system disorders) | 1
Multi-Organ Failure (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Skin And Subcutaneous Tissue Disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 1
Treatment Related Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BRAF (Dabrafenib) and MEK (Trametinib) Inhibitors (N=17)
Abdominal Pain (Gastrointestinal disorders) | 4
Alanine Aminotransferase Increased (Investigations) | 13
Alkaline Phosphatase Increased (Investigations) | 4
Allergic Reaction (Immune system disorders) | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Anemia (Blood and lymphatic system disorders) | 11
Anorexia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Aspartate Aminotransferase Increased (Investigations) | 13
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Blood Bilirubin Increased (Investigations) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Cataract (Eye disorders) | 1
Chills (General disorders) | 11
Chronic Kidney Disease (Renal and urinary disorders) | 1
Confusion (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Cpk Increased (Investigations) | 2
Creatinine Increased (Investigations) | 6
Dehydration (Metabolism and nutrition disorders) | 2
Depression (Psychiatric disorders) | 2
Diarrhea (Gastrointestinal disorders) | 10
Dizziness (Nervous system disorders) | 5
Dry Mouth (Gastrointestinal disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 4
Dysgeusia (Nervous system disorders) | 1
Dysmenorrhea (Reproductive system and breast disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Edema Face (General disorders) | 1
Edema Limbs (General disorders) | 5
Ejection Fraction Decreased (Investigations) | 2
Endocrine Disorders - Other, Specify (Endocrine disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1
Eye Disorders - Other, Specify (Eye disorders) | 3
Eye Pain (Eye disorders) | 1
Fatigue (General disorders) | 13
Fever (General disorders) | 12
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Floaters (Eye disorders) | 1
Flu Like Symptoms (General disorders) | 8
Flushing (Vascular disorders) | 2
Fracture (Injury, poisoning and procedural complications) | 1
Gait Disturbance (General disorders) | 1
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2
Gastrointestinal Disorders - Other, Specify (Gastrointestinal disorders) | 4
General Disorders And Administration Site Conditions - Other, Specify (General disorders) | 3
Generalized Muscle Weakness (General disorders) | 2
Ggt Increased (Investigations) | 4
Gum Infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 8
Hemorrhoids (Gastrointestinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hot Flashes (Vascular disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 7
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 7
Hyperthyroidism (Endocrine disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 13
Hypocalcemia (Metabolism and nutrition disorders) | 8
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hypotension (Vascular disorders) | 2
Hypothyroidism (Endocrine disorders) | 2
Infections And Infestations - Other, Specify (Infections and infestations) | 1
Insomnia (Psychiatric disorders) | 1
Intracranial Hemorrhage (Nervous system disorders) | 1
Libido Decreased (Psychiatric disorders) | 1
Lipase Increased (Investigations) | 2
Lymphocyte Count Decreased (Investigations) | 16
Lymphocyte Count Increased (Investigations) | 1
Malaise (General disorders) | 3
Memory Impairment (Nervous system disorders) | 1
Musculoskeletal And Connective Tissue Disorder - Other, Specify (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Nail Loss (Skin and subcutaneous tissue disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3
Nausea (Gastrointestinal disorders) | 10
Neck Pain (Musculoskeletal and connective tissue disorders) | 3
Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps) - (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neutrophil Count Decreased (Investigations) | 10
Non-Cardiac Chest Pain (General disorders) | 2
Pain (General disorders) | 5
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2
Pain Of Skin (Skin and subcutaneous tissue disorders) | 3
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1
Papulopustular Rash (Infections and infestations) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Personality Change (Psychiatric disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Platelet Count Decreased (Investigations) | 9
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5
Psychiatric Disorders - Other, Specify (Psychiatric disorders) | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 9
Reproductive System And Breast Disorders - Other, Specify (Reproductive system and breast disorders) | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, Thoracic And Mediastinal Disorders - Other, Specify (Respiratory, thoracic and mediastinal disorders) | 1
Seizure (Nervous system disorders) | 1
Sinus Pain (Nervous system disorders) | 2
Sinusitis (Infections and infestations) | 2
Skin And Subcutaneous Tissue Disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 13
Skin Induration (Skin and subcutaneous tissue disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3
Stomach Pain (Gastrointestinal disorders) | 2
Tooth Infection (Infections and infestations) | 1
Tremor (Nervous system disorders) | 1
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2
Urinary Incontinence (Renal and urinary disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1
Urinary Tract Pain (Renal and urinary disorders) | 2
Vaginal Infection (Infections and infestations) | 1
Vaginal Pain (Reproductive system and breast disorders) | 2
Vomiting (Gastrointestinal disorders) | 9
Watering Eyes (Eye disorders) | 1
Weight Gain (Investigations) | 1
Weight Loss (Investigations) | 2
White Blood Cell Decreased (Investigations) | 13
Wound Infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT01726738/Prot_SAP_000.pdf